CLINICAL TRIAL: NCT06088303
Title: Enhancing PTSD Treatment Outcomes by Improving Patient-Provider Communication
Acronym: AWARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-44384; 1K23MH132815-01A1 (NIH)
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Posttraumatic stress disorder; Cognitive processing therapy; Prolonged exposure; Adjunctive writing for amplifying response and engagement; Health communication; Patient-provider communication
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPT/PE with AWARE (Experimental): Participants randomized into this arm will receive either cognitive processing therapy (CPT) or prolonged exposure (PE) with the adjunctive writing intervention to amplify response and engagement (AWARE).
  CPT and PE are both recommended as gold standard treatments by published PTSD clinical practice guidelines. Participants will choose whether to receive CPT or PE. The standard treatment length will be 8-15 weekly sessions; however, participants and providers may collaboratively agree to early completion or additional sessions as warranted. AWARE will be integrated into the CPT/PE sessions.
  Interventions: Behavioral: Adjunctive writing to amplify response and engagement (AWARE); Behavioral: Cognitive processing therapy (CPT); Behavioral: Prolonged exposure (PE)
- CPT/PE TAU (Active Comparator): Participants randomized into this arm will receive either cognitive processing therapy (CPT) or prolonged exposure (PE) treatment as usual (TAU).
  CPT and PE are both recommended as gold standard treatments by published PTSD clinical practice guidelines. Participants will choose whether to receive CPT or PE. The standard treatment length will be 8-15 weekly sessions; however, participants and providers may collaboratively agree to early completion or additional sessions as warranted.
  Interventions: Behavioral: Cognitive processing therapy (CPT); Behavioral: Prolonged exposure (PE)

INTERVENTIONS:
Behavioral: Adjunctive writing to amplify response and engagement (AWARE) — AWARE includes two components: 1) patients complete brief writing prompts asking about their experiences in treatment, and 2) therapists review patients' responses and facilitate guided discussion related to patients' experiences during check-ins at the beginning of each session.
  Arms: CPT/PE with AWARE
Behavioral: Cognitive processing therapy (CPT) — CPT is a manualized, evidence-based therapy for PTSD typically delivered over the course of 8-15 weekly 60-minute sessions. CPT focuses on helping patients identify trauma-related stuck points (inaccurate and/or unhelpful beliefs) and challenge those beliefs to arrive at healthier, more balanced beliefs about their traumatic experiences, themselves, others, and the world.
Behavioral: Prolonged exposure (PE) — PE is a manualized, evidence-based therapy for PTSD typically delivered over the course of 8-15 weekly 90-minute sessions. PE focuses on reducing unhelpful avoidance and helping patients process and make sense of their traumatic experiences through in vivo and imaginal exposure to trauma-related reminders and memories.

SUMMARY:
The purpose of this clinical trial is to learn whether existing treatments for posttraumatic stress disorder (PTSD) can be improved. Two treatments for PTSD, cognitive processing therapy (CPT) and prolonged exposure (PE) will be studied. CPT and PE are effective treatments that are widely available, but interventions are needed to improve patient outcomes in these treatments. The investigators have developed an Adjunctive Writing intervention for Amplifying Response and Engagement (AWARE), which was designed using health communication strategies to enhance CPT and PE by improving communication between patients and therapists about patients' experiences in treatment. This research will investigate whether adding AWARE to CPT and PE will lead to better treatment outcomes compared to CPT and PE provided as usual without AWARE. AWARE includes a brief writing task asking patients about their experiences in treatment, as well as guided therapist responses to improve patient-therapist communication about patients' experiences in treatment. In the first phase of the study (case series phase), CPT or PE with AWARE will be provided to four adults with PTSD to pilot test adding AWARE to CPT and PE, seek patient and provider feedback, and refine AWARE. The first four participants who enroll will be part of the case series and will receive CPT or PE with AWARE. Then, in the second phase of the study, the randomized controlled trial (RCT) phase, the investigators will enroll 50 more adults with PTSD who will be randomly assigned (like flipping a coin) to receive CPT/PE as usual or CPT/PE with AWARE. It is expected that 25 participants will be randomized to CPT/PE with AWARE and 25 participants will be randomized to receive CPT/PE provided as usual. The goals of the RCT phase are to study whether AWARE is acceptable to patients, whether it is feasible to add AWARE to CPT and PE, and whether adding AWARE to CPT and PE improves patient-therapist communication and treatment outcomes compared to CPT/PE as usual.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD
* Stable on psychiatric medications for at least 4 weeks

Exclusion Criteria:

* Current unstable bipolar disorder
* Current psychosis
* Current active suicidal or homicidal ideation with intent or plan
* Current severe substance use that warrants immediate medical attention
* Current trauma-focused treatment
* Significant cognitive impairment that would prevent engagement in assessments and therapy (e.g., advanced dementia, severe traumatic brain injury).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-provider communication: VR-CoDES (Posttreatment) | Immediately after ending treatment
  Verona Coding Definitions of Emotional Sequences (VR-CoDES) - Observational Coding - Used to code patient writing and recordings of each weekly session check-in for 1) patient disclosure of concerns and 2) therapists' responses to patients' concerns. A random selection of 25% of session recordings will be rated. Patients' cues and concerns and providers' responses to patients' cues and concerns are classified into 25 categories, coded as present/absent. Codes will be averaged across all treatment sessions coded.
PTSD: CAPS-5 (Posttreatment) | Immediately after ending treatment
  Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 (CAPS-5) - Clinician Interview - The CAPS-5 includes 20 items assessing PTSD symptom severity. Total scores range from 0-80 with higher scores indicating more severe PTSD symptoms.
PTSD: CAPS-5 (Follow-up) | 3 months after ending treatment
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) - Clinician Interview - The CAPS-5 includes 20 items assessing PTSD symptom severity. Total scores range from 0-80 with higher scores indicating more severe PTSD symptoms.
Feasibility assessed by CPT adherence | Immediately after ending treatment
  CPT Therapist Adherence and Competence Protocol-Revised - Observer Rating - CPT adherence is the percentage of CPT protocol elements completed across therapy sessions, rated from 0-100%, with a higher percentage indicating greater adherence. A random selection of 50% of session recordings will be rated, and ratings will be averaged across all rated sessions. Completion of ≥ 90% mean adherence to protocol elements indicates high CPT adherence, and would be an indicator of feasibility of AWARE.
Feasibility assessed by CPT competence | Immediately after ending treatment
  CPT Therapist Adherence and Competence Protocol-Revised - Observer Rating - CPT competence is the skill with which therapists implement CPT protocol elements across therapy sessions, rated from 1-7, with higher scores indicating greater competence. A random selection of 50% of session recordings will be rated, and ratings will be averaged across all rated sessions. A score of good (5) or greater on the 1-7 scale indicates high CPT competence, and would be an indicator of feasibility of AWARE.
Feasibility assessed by PE adherence | Immediately after ending treatment
  PE Fidelity Rating Form - Observer Rating - PE adherence is the percentage of PE protocol elements completed across therapy sessions, rated from 0-100%, with a higher percentage indicating greater adherence. A random selection of 50% of session recordings will be rated, and ratings will be averaged across all rated sessions. Completion of ≥ 90% mean adherence to protocol elements indicates high PE adherence, and would be an indicator of feasibility of AWARE.
Feasibility assessed by PE competence | Immediately after ending treatment
  PE Fidelity Rating Form - Observer Rating - PE competence is the skill with which therapists implement PE protocol elements across therapy sessions, rated from 1-7, with higher scores indicating greater competence. A random selection of 50% of session recordings will be rated, and ratings will be averaged across all rated sessions. A score of good (5) or greater on the 1-7 scale indicates high PE competence, and would be an indicator of feasibility of AWARE.
Acceptability: Client satisfaction (Mid-treatment) | After 6 sessions
  Client Satisfaction Questionnaire (CSQ) - Self-Report - The CSQ has 8 items assessing client satisfaction with the treatment they have received. Total scores range from 8-32; higher scores indicate greater client satisfaction/treatment acceptability.
Acceptability: Client satisfaction (Posttreatment) | Immediately after ending treatment
  Client Satisfaction Questionnaire (CSQ) - Self-Report - The CSQ has 8 items assessing client satisfaction with the treatment they have received. Total scores range from 8-32; higher scores indicate greater client satisfaction/treatment acceptability.
Acceptability: Therapeutic Alliance (Mid-treatment) | After 6 sessions
  Working Alliance Inventory Short-Revised (WAI-SR) - Self-Report - The WAI-SR has 12 items assessing three aspects of the therapeutic alliance: agreement on tasks, agreement on goals, and therapeutic bond. Total scores range from 12-60; higher scores indicate stronger therapeutic alliance/treatment acceptability.
Acceptability: Therapeutic Alliance (Posttreatment) | Immediately after ending treatment
  Working Alliance Inventory Short-Revised (WAI-SR) - Self-Report - The WAI-SR has 12 items assessing three aspects of the therapeutic alliance: agreement on tasks, agreement on goals, and therapeutic bond. Total scores range from 12-60; higher scores indicate stronger therapeutic alliance/treatment acceptability.
Treatment Completion | Immediately after ending treatment
  Proportion of patients who completed a full course of the assigned treatment

SECONDARY OUTCOMES:
Patient-provider communication: PPIS (Posttreatment) | Immediately after ending treatment
  Patient-Provider Interaction Scale (PPIS) - Self-Report - The PPIS has 6 items assessing patients' perceptions of patient-provider communication. The PPIS will be collected every session by study staff, and scores will be averaged across sessions. Total scores range from 6-24; higher scores indicate better patient-provider communication.
PTSD: PCL-5 (Posttreatment) | Immediately after ending treatment
  PTSD Checklist for DSM-5 (PCL-5) - Self-Report - The PCL-5 has 20 items assessing PTSD symptom severity. Total scores range from 0-80 with higher scores indicating more severe PTSD symptoms.
PTSD: PCL-5 (Follow-up) | 3 months after ending treatment
  PTSD Checklist for DSM-5 (PCL-5) - Self-Report - The PCL-5 has 20 items assessing PTSD symptom severity. Total scores range from 0-80 with higher scores indicating more severe PTSD symptoms.
Depression (Posttreatment) | Immediately after ending treatment
  Patient Health Questionnaire (PHQ-9) - Self-Report - The PHQ-9 has 9 items assessing depression symptoms. Total scores range from 0-27; higher scores indicating greater depression severity.
Depression (Follow-Up) | 3 months after ending treatment
  Patient Health Questionnaire (PHQ-9) - Self-Report - The PHQ-9 has 9 items assessing depression symptoms. Total scores range from 0-27; higher scores indicating greater depression severity.
Functional impairment (Posttreatment) | Immediately after ending treatment
  World Health Organization Disability Assessment Schedule-II (WHODAS-II) - Self-Report - The WHODAS-II has 36 items assessing disability and functional impairment. Total scores range from 0-144; higher scores indicate greater disability/functional impairment.
Functional impairment (Follow-up) | 3 months after ending treatment
  World Health Organization Disability Assessment Schedule-II (WHODAS-II) - Self-Report - The WHODAS-II has 36 items assessing disability and functional impairment. Total scores range from 0-144; higher scores indicate greater disability/functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Alpert, PhD, Principal Investigator — National Center for PTSD at VA Boston Healthcare System, BU School of Medicine, Psychiatry
Locations (1):
- National Center for PTSD at VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified demographic and raw quantitative data will be deposited into the NIMH Data Archive (NDA). All data will be de-identified prior to receipt by the repository. Data will be de-identified pursuant to the HIPAA Privacy Rule, 45 CFR § 164.514(b). A brief study protocol will also be submitted to NDA and will be made freely available.
Supporting Information: Study Protocol
Time Frame: Data will be deposited starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates. Data generated from this project will be made available as soon as possible, and no later than the time of publication or the end of the funding period, whichever comes first. The duration of preservation and sharing of the data is controlled by the NDA; NDA currently has no process for deleting or retiring datasets, and thus far no data has been removed to our knowledge.
Access Criteria: To request access to the data, researchers can use the standard processes at NDA; the NDA Data Access Committee will review requests and decide which requests to grant. The standard NDA access process allows access for one year and is renewable thereafter.